CLINICAL TRIAL: NCT06988046
Title: Clinical Effects of an Innovative Three-Dimensional Orthosis in Thoracic Hyperkyphosis: A Randomized Controlled Trial
Brief Title: Innovative Orthosis in Hyperkyphosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, sena ozdemir, PhD, PT, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: E-30 10840098-772.02-6671
Record Dates: First submitted 2025-05-16; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2021-12

CONDITIONS: Postural Kyphosis; Hyperkyphosis
Keywords: Thoracic hyperkyphosis; postural kyphosis; three-dimensional orthosis; thoracic kyphosis angle
MeSH Terms: conditions — Kyphosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cover spine orthosis group (CSO) (Experimental): he Cover Spine Orthosis (CSO) is a novel therapeutic device specifically engineered to address excessive thoracic curvature in individuals diagnosed with hyperkyphosis. Utilizing three-dimensional (3D) printing technology, the orthosis is produced from thermoplastic polyurethane, a material known for its flexibility and durability. The CSO incorporates two primary corrective components positioned anteriorly and posteriorly. The anterior section functions to stabilize the thoracic region from the front, while the posterior section delivers a corrective force from the back, targeting spinal alignment. To ensure a secure and adaptive fit, elastic webbing with Velcro and loop fasteners is integrated on both sides of the shoulder and trunk. These connectors link the anterior and posterior components, maintaining optimal suspension of the orthosis on the user's body. Furthermore, the design features a broad contact area, which enhances postural control by distributing mechanical forces more
  Interventions: Device: Cover spine orthosis (CSO)
- Semi-rigid thoracolumbar orthosis group (SRTLO) (Active Comparator): The control group was fitted with a semi-rigid thoracolumbar orthosis (SRTLO), a device whose clinical efficacy has been previously validated. This orthosis includes paraspinal support bars, bilateral shoulder straps, and a Velcro-based fastening system. The paraspinal bars function to limit spinal flexion, thereby promoting an extended spinal posture. The shoulder straps are passed anteriorly over the shoulders, routed posteriorly through the axillary regions, crossed to the opposite side, and brought back to the front. Once appropriate tension is applied, the straps are secured using Velcro fasteners. Final stabilization is accomplished by anterior traction on the thoracic section straps to ensure optimal corrective force distribution.
  Interventions: Device: Semi-rigid thoracolumbar orthosis

INTERVENTIONS:
Device: Cover spine orthosis (CSO) — The participants included in the study were asked to use the orthoses given as a result of randomization for four weeks, excluding the time they were asleep (average 12 h per day).
  Arms: Cover spine orthosis group (CSO)
Device: Semi-rigid thoracolumbar orthosis — The participants included in the study were asked to use the orthoses given as a result of randomization for four weeks, excluding the time they were asleep (average 12 h per day).
  Arms: Semi-rigid thoracolumbar orthosis group (SRTLO)

SUMMARY:
Thoracic hyperkyphosis is a common postural deformity; however, the optimal treatment strategy has yet to be clearly defined. This randomized controlled trial aimed to assess the effectiveness of an innovative three-dimensional printed Cover Spine Orthosis (CSO) in managing thoracic hyperkyphosis. Specifically, the study compared the effects of the CSO on kyphosis angle, quality of life (QoL), and user satisfaction with those of a semi-rigid thoracolumbar orthosis (SRTLO) that has established efficacy in the literature.

DETAILED DESCRIPTION:
Postural kyphosis is associated with various clinical symptoms, including fatigue, pain, weakness of the back extensor muscles, depressive mood, and a reduction in quality of life (QoL). Previous research has consistently shown that spinal deformities negatively impact overall health, particularly diminishing individuals' QoL. Although conservative approaches are commonly recommended for managing postural kyphosis, a universally accepted treatment protocol has not yet been established. Current evidence suggests that interventions such as exercise, kinesio-taping, and orthotic use may be effective in decreasing the thoracic kyphosis angle (TKA). Among these, orthotic interventions have been widely employed to correct posture and reduce TKA. While various orthosis designs have been studied, and some have demonstrated significant outcomes, there is still no consensus on the most effective orthotic treatment. In light of existing literature and advancements in biomechanics and design technologies, a novel three-dimensional (3D) orthosis was developed to address these gaps. This study aimed primarily to assess the effectiveness of a custom-designed, 3D-printed Cover Spine Orthosis (CSO) in reducing TKA in individuals with postural kyphosis, in comparison to a semi-rigid thoracolumbar orthosis (SRTLO) previously validated in the literature. A secondary objective was to evaluate and compare the effects of both orthoses on quality of life and user satisfaction

ELIGIBILITY:
Inclusion Criteria:

* Individuals of both sexes (male and female)
* Aged between 20 and 60 years
* Presence of thoracic kyphosis angle (TKA) ≥ 40°

Exclusion Criteria:

* History of spinal surgery or traumatic injury
* Received physiotherapy treatment within the last six months
* Diagnosed with congenital spinal deformities or scoliosis
* Presence of acute musculoskeletal injury
* Inability to tolerate or adapt to orthotic application

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Thoracic kyphosis angle (TKA) | 3 minutes
  Thoracic kyphosis angle (TKA) was assessed using a flexicurve, a flexible, plastic-coated metal ruler that conforms to the curvature of the spine. For measurement, the flexicurve was molded along the thoracic spine between the C7 and T12 vertebrae while the participant maintained an upright posture. Once the curve was shaped, its outline was transferred onto paper for further analysis. The kyphosis index was calculated by measuring the height of the apex of the curve (B) and dividing it by the total horizontal length of the thoracic curve (X), then multiplying the result by 100: (B/X) × 100. Additionally, the flexicurve angle (θ) was derived by constructing a triangle from the traced curve and measuring the angle formed by lines drawn perpendicular to its sides.

SECONDARY OUTCOMES:
Quality of life (QoL) | 3 minutes
  Participant quality of life (QoL) was assessed using the Scoliosis Research Society-22 (SRS-22) questionnaire. This instrument comprises 22 items divided into five distinct domains: pain, self-image, spinal function, mental health, and satisfaction with treatment. Each item is scored on a 5-point likert scale ranging from 1 (least favorable) to 5 (most favorable). Higher total and subscale scores reflect better perceived quality of life, whereas lower scores indicate reduced well-being.
User satisfaction | 2 minutes
  User satisfaction was measured using the Quebec User Evaluation of Satisfaction with Assistive Technology 2.0 (QUEST 2.0), a validated instrument designed to assess satisfaction with assistive technologies. The questionnaire consists of 12 items divided into two subdomains: device-related (8 items) and service-related (4 items). These items evaluate features such as size, weight, usability, comfort, and overall effectiveness. Responses are rated on a 5-point Likert scale, ranging from 1 (not satisfied at all) to 5 (very satisfied), with higher scores reflecting greater satisfaction with the device or service.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University Prosthetics-Orthotics Research Center (POMER), Istanbul, Kavacık, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The datasets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request.

REFERENCES:
- See also: Related Info — https://journals.lww.com/md-journal/fulltext/2025/03210/effect_of_digital_health_corrective_posture.66.aspx